CLINICAL TRIAL: NCT01977183
Title: Effects of MSPrebiotic on Gut Health in the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Boniface Hospital (Other)
Collaborators: National Microbiology Laboratory, Canada (Other); MSP Starch Products Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RRC/2013/1285; B2013:016 (Other: University of Manitoba Biomedical Reserach Ethics Board)
Record Dates: First submitted 2013-10-11; First posted 2013-11-06 (Estimated); Last update posted 2023-01-06 (Actual); Status verified 2015-07

CONDITIONS: Focus of Study; Impact of MSPrebiotic on Gastrointestinal Microbiota
Keywords: gastrointestinal; microbiome; prebiotic; starch

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Elderly adults with MSPrebiotic (Experimental): 30 g of MSPrebiotic (potato resistant starch) per day taken with 1 glass (approximately 250 mL) of non-heated fluid or non-heated semi-solid food. If the participant is taking any medications, they will be advised to either take the product 2 hours before or 2 hours after any medications.
  Interventions: Dietary Supplement: MSPrebiotic
- Elderly adults with Placebo (Placebo Comparator): 30 g of corn starch per day taken with 1 glass (approximately 250 mL) of non-heated fluid or or non-heated semi-solid food. If the participant is taking any medications, they will be advised to either take the product 2 hours before or 2 hours after any medications.
  Interventions: Dietary Supplement: Placebo
- General adult population with MSPrebiotic (Experimental): 30 g of MSPrebiotic (potato resistant starch) per day taken with 1 glass (approximately 250 mL) of non-heated fluid. If the participant is taking any medications, they will be advised to either take the product 2 hours before or 2 hours after any medications.
  Interventions: Dietary Supplement: MSPrebiotic
- General adult population with Placebo (Placebo Comparator): 30 g of corn starch per day taken with 1 glass (approximately 250 mL) of non-heated fluid. If the participant is taking any medications, they will be advised to either take the product 2 hours before or 2 hours after any medications.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: MSPrebiotic — Potato Resistant Starch
  Other Names: Potato Resistant Starch
  Arms: Elderly adults with MSPrebiotic; General adult population with MSPrebiotic
Dietary Supplement: Placebo — Placebo - Corn Starch
  Arms: Elderly adults with Placebo; General adult population with Placebo

SUMMARY:
The purpose of this clinical trial is to study the effects of potato resistant starch on the microbiota (microorganisms or bacteria) and short chain fatty acids levels of the gut. Levels will be measured and compared between elderly adults and in pre-elderly, adults from the general public. A correlation between the use of potato resistant starch and specific clinical and quality of life endpoints between elderly adults and in pre-elderly, adults from the general public will be studied.

Hypothesis 1: The investigator hypothesizes that the microbiome in elderly adults (≥70 years) is less diverse and more prone to imbalance compared to adults (30-50 years) from the general population and that this imbalance of the gut microflora in the elderly adults is partially related to inadequate RS in their diet.

Hypothesis 2: The investigator hypothesizes that ingestion of potato resistant starch of food grade quality (MSPrebiotic) will stabilize the gut microbiome (i.e. high Firmicutes/Bacteroides ratio)in LTC residents (i.e. similar to that of adults from the general population), thereby improving gut health and reducing the risk of diarrhea and/or gut infection.

DETAILED DESCRIPTION:
To assess the impact on the potato resistant starch on the microbiota, pyrosequencing will be performed on stool samples to determine the original composition and assess any changes over the study period. In addition the impact of the potato resistant starch on inflammatory markers will be assess through blood samples collected over the study period.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent
* Willing to provide stool and blood specimens 5 times over the 14 week study period
* Subjects ≥ 70 years of age
* Subjects 30-50 years of age

Exclusion Criteria:

* Pregnancy
* Crohn's disease or any other inflammatory bowel disease
* Individuals with Lupus, or on cancer chemotherapy
* Pre-diabetes or Diabetes
* Thyroid disease
* Renal disease
* Hepatic disease
* Previous gastrointestinal surgery (intestinal resection, gastric bypass, colorectal surgery)
* Subjects on probiotic
* Subjects on antibiotics at time of recruitment or on antibiotics within the previous five weeks
* Individuals experiencing dysphagia
* Subjects using additional fiber supplements
* Subjects on digestants, emetics and antiemetics, medications for acid peptic disease and antacids.

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2013-09; Primary Completion 2016-01 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Tolerability of 30g dose of MSPrebiotic | 2, 6, 10 and 14 weeks
  Changes from baseline in the tolerability of ingestion of 30 g once/day of MSPrebiotic with respect to gastrointestinal side effects (excessive flatulence, changes in bowel movements, abdominal pain and bloating) at 2, 6, 10 and 14 weeks.
Gut health improvements | 2, 6, 10 and 14 weeks
  Changes from baseline in gut health improvements including: reduced constipation (i.e. improved ease of bowel movements without stool softeners), microbiome composition (i.e. favourable Firmicutes to Bacteroides ratio) at 2, 6, 10 and 14 weeks.
Levels of short chain fatty acids in stool and lipid level in blood | 2, 4, 6, 10 and 14 weeks
  Changes from baseline of short chain fatty acid levels in stool including; acetate, propionate, butyrate, isobutyrate, valerate, isovalerate at 2, 4, 6, 10 and 14 weeks.
Inflammatory marker | 2, 6, 10 and 14 weeks
  Changes from baseline of Inflammatory marker (IL-10, C-reactive protein, TNFα) levels in blood at 2, 6, 10 and 14 weeks.

SECONDARY OUTCOMES:
Changes from baseline in overall health at 2, 6, 10 and 14 weeks | 2, 6, 10 and 14 weeks
  This will be assessed based on completion of a daily health log that assesses a wide variety of parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle J Alfa, PhD, Principal Investigator — St. Boniface Hospital Research Centre
Locations (2):
- Canada (2):
  - St. Boniface Hosptial Research Centre, Winnipeg, Manitoba
  - Deer Lodge Centre, Winnipeg, Manitoba

REFERENCES:
- [Derived] Bush JR, Alfa MJ. Increasing levels of Parasutterella in the gut microbiome correlate with improving low-density lipoprotein levels in healthy adults consuming resistant potato starch during a randomised trial. BMC Nutr. 2020 Dec 11;6(1):72. doi: 10.1186/s40795-020-00398-9. PMID 33303023
- [Derived] Alfa MJ, Strang D, Tappia PS, Olson N, DeGagne P, Bray D, Murray BL, Hiebert B. A Randomized Placebo Controlled Clinical Trial to Determine the Impact of Digestion Resistant Starch MSPrebiotic(R) on Glucose, Insulin, and Insulin Resistance in Elderly and Mid-Age Adults. Front Med (Lausanne). 2018 Jan 22;4:260. doi: 10.3389/fmed.2017.00260. eCollection 2017. PMID 29410955
- [Derived] Alfa MJ, Strang D, Tappia PS, Graham M, Van Domselaar G, Forbes JD, Laminman V, Olson N, DeGagne P, Bray D, Murray BL, Dufault B, Lix LM. A randomized trial to determine the impact of a digestion resistant starch composition on the gut microbiome in older and mid-age adults. Clin Nutr. 2018 Jun;37(3):797-807. doi: 10.1016/j.clnu.2017.03.025. Epub 2017 Mar 31. PMID 28410921